CLINICAL TRIAL: NCT04455867
Title: The Sunnybrook Type 2 Diabetes Study
Acronym: S2DS
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Walter Swardfager, Principal Investigator, Sunnybrook Health Sciences Centre
Other Study IDs: 422-2015; 0939 (Registry Identifier: Clinical Trials Ontario)
Record Dates: First submitted 2020-06-22; First posted 2020-07-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; PreDiabetes
Keywords: Mood; Cognition; Brain Imaging; Type 2 Diabetes; Sleep; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Motor Activity | interventions — Ambulatory Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Serum Plasma White blood cells Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UHN Toronto Rehab: Participants with prediabetes of T2DM undertaking a 6-month stepped hybrid (home and clinic based) aerobic plus resistance exercise intervention as per the site's standard protocol (Diabetes Exercise and Healthy Lifestyle Program).
  Interventions: Behavioral: Diabetes Exercise and Healthy Lifestyle Program
- Sunnybrook Health Sciences Centre: Participants with prediabetes or T2DM receiving care from an outpatient service at Sunnybrook Health Sciences Centre.
  Interventions: Other: Outpatient care

INTERVENTIONS:
Behavioral: Diabetes Exercise and Healthy Lifestyle Program — The program combines exercise, education and healthy lifestyle behaviour changes. Participants will begin the program with a cardiopulmonary exercise assessment. Then the team will create a personalized program of exercise based on functional abilities and personal goals. Participants will attend 1 supervised exercise class a week, which includes a warm-up and stretching routine, aerobic exercise (walking, stationary cycling or elliptical machine), resistance training and an educational session. This program also offers peer-to-peer support and encourages participants to carry out their own exercise program at home 4 more times per week and to keep a weekly exercise diary to help them with their progress.
  Groups: UHN Toronto Rehab
Other: Outpatient care — Participants receive usual care from outpatient services, which may include Endocrinology, Family Medicine, or Diabetes Education
  Groups: Sunnybrook Health Sciences Centre

SUMMARY:
The Sunnybrook Type 2 Diabetes Study (S2DS) is a prospective observational study of people with prediabetes or Type 2 Diabetes Mellitus (T2DM), that aims to understand the aetiologies, manifestations, and clinical consequences of mood and cognitive complications. The study recruits from the services at Sunnybrook Health Sciences Centre and from the neighbouring University Health Network Toronto Rehabilitation Institute Cardiac Rehabilitation Program.

DETAILED DESCRIPTION:
The S2DS is a prospective observational study of people with prediabetes or T2DM recruited from Sunnybrook Health Sciences Centre and the neighbouring University Health Network Toronto Rehabilitation Institute Cardiac Rehabilitation Program. Participants recruited from Sunnybrook are receiving care from services there (e.g. Family Medicine, Endocrinology, and the Sunnybrook Diabetes Education Centre). Participants recruited from the Toronto Rehab are undertaking a 6-month stepped hybrid (home and clinic based) aerobic plus resistance exercise intervention as part of a program at that site (e.g. the Diabetes, Exercise, and Healthy Lifestyle Program).

Study assessments are conducted at baseline, 3 months, 6 months and 18 months. Main outcomes include cognitive performance, assessed using a detailed neurocognitive battery, and mood symptoms assessed via research criteria for a depressive episode and self-report instruments. Other lifestyle factors are also examined, including physical activity, sleep quality, diet, and subjective stress. Diabetes complications and characteristics are monitored, as are all concomitant medications and supplements. With permission, participant data are linked prospectively to public health records to ascertain long-term outcomes and health services utilization.

The cohort is characterized using biological, neuroimaging and biometric measures. Fasting morning blood and urine samples are taken at each assessment. Serum, plasma, whole blood, and white blood cells are bio-banked for biochemical, genetic and other analyses. The MRI study includes a 1.5 hr MRI scan at 3.0 T. Sequences performed include structural imaging (T1, T2, DTI and FLAIR) and resting state functional MRI. Two optional sub-studies are offered: a cerebrovascular reactivity MRI protocol, and a sleep quality and apnea protocol (baseline, 6 month and 18 month visits). The sleep study uses an overnight wearable sleep monitor.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one of the following: high HbA1c, impaired fasting glucose (IFG), impaired glucose tolerance (IGT), but not yet diagnosed with Type 2 diabetes or have a diagnosis of Type 2 diabetes.
* Be able to communicate in English
* Be 18 years of age or older

Exclusion Criteria:

* Pregnancy
* Inability to give informed consent
* Current cancer diagnosis
* Have a prior diagnosis of bipolar disorder or schizophrenia.
* Have a prior diagnosis of a neurological and/or neurodegenerative disorder.
* Have a current substance use disorder or a previous substance use disorder diagnosed within the last 5 years (excluding nicotine)
* Poor score on the Mini Mental State Examination (MMSE)

Exclusion criteria (Brain Imaging Sub-Study):

* Contraindications to SHSC's MRI safety protocol.
* Participants that do not meet the inclusion/exclusion criteria of the main study.

Exclusion criteria for (Brain Imaging Sub-Study - CVR procedure):

* Use of medical equipment that would interfere with the placement of the CVR mask.
* Significant pulmonary disease (e.g. asthma, pulmonary fibrosis, emphysema, chronic obstructive pulmonary disease, pulmonary vascular disease, pleural disorders, pneumonia)
* Participants that do not meet the criteria for the MRI sub-study.

Exclusion criteria (Sleep Quality and Apnea Sub-Study):

* Participants that have a medical device that would interfere with placement of portable sleep monitor equipment i.e. Participant requires O2 therapy and uses nasal prongs
* Participants that have a condition that may compromise accuracy of the HSAT results i.e. moderate-severe pulmonary disease or congestive heart failure
* Participants that do not meet the inclusion/exclusion criteria of the main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals with prediabetes or T2DM who are receiving care from an outpatient service at Sunnybrook Health Sciences Centre, or as part of the Diabetes and Healthy Lifestyle Program at the University Health Network Toronto Rehabilitation Institute Cardiac Rehabilitation Program.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Depressive episode | 6 Months
  Depressive episodes are identified using a Structured Clinical Interview for the DSM-5 criteria (SCID-5RV).
Neuropsychological function | 6 Months
  A Z-score computed from a sensitive neuropsychological battery is administered based on the Canadian Stroke Network & National Institutes of Neurological Disorders recommendations.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, 3 Month, 6 Month, 18 Month
  Depressive symptoms are monitored using the Beck Depression Inventory-II (BDI-II).
Cognitive Status | Baseline, 3 Month, 6 Month, 18 Month
  Cognitive status is monitored using the Montreal Cognitive Assessment (MoCA).

CONTACTS AND LOCATIONS:
Overall Officials: Walter Swardfager, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anita NZ, Forkan N, Kamal R, Nguyen MM, Yu D, Major-Orfao C, Wong SK, Lanctot KL, Herrmann N, Oh PI, Shah BR, Gilbert J, Assal A, Halperin IJ, Pedersen TL, Taha AY, Swardfager W. Serum soluble epoxide hydrolase related oxylipins and major depression in patients with type 2 diabetes. Psychoneuroendocrinology. 2021 Apr;126:105149. doi: 10.1016/j.psyneuen.2021.105149. Epub 2021 Jan 19. PMID 33503568